CLINICAL TRIAL: NCT06620679
Title: Mapping the Effect of (neuro)inflammation on Stress Sensitivity in the Brain of Healthy Men
Acronym: INFLAMES
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Principal Investigator, Lukas Van Oudenhove, Principal Investigator, Universitaire Ziekenhuizen KU Leuven
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: S67872; 101002525 (Other Grant/Funding Number: ERC Consolidator Grant)
Record Dates: First submitted 2024-09-24; First posted 2024-10-01 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Inflammation; Stress; Healthy Volunteer
Keywords: Inflammation; Stress; Lipopolysaccharide (LPS); Short-chain fatty acids; Neuroimaging
MeSH Terms: conditions — Inflammation | interventions — Lipopolysaccharides

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- LPS then Saline (Experimental): A crossover arm where the participant first receives the intervention (LPS), undergoes a wash-out period, then receives the placebo (saline).
  Interventions: Biological: Lipopolysaccharide (LPS); Other: Placebo
- Saline then LPS (Experimental): A crossover arm where the participant first receives the placebo (saline), undergoes a wash-out period, then receives the intervention (LPS).
  Interventions: Biological: Lipopolysaccharide (LPS); Other: Placebo

INTERVENTIONS:
Biological: Lipopolysaccharide (LPS) — Lipopolysaccharide (LPS), single i.v. bolus, 0.4 ng/kg body weight
Other: Placebo — Normal saline, single i.v. bolus, in equal volume to intervention

SUMMARY:
The goal of this interventional study is to determine the effects of inflammation on stress responses in the brain of healthy men. In order to achieve this goal, participants are injected with an inflammation-inducing agent, then observed inside a brain scanner.

DETAILED DESCRIPTION:
This interventional study is a randomized, triple-blind, placebo-controlled, cross-over study aiming to elucidate the impact of acute laboratory-induced inflammation using lipopolysaccharide (LPS) on stress responses in the brain of healthy men. Acute stress responses to a psychological task, the Maastricht Imaging Stress Task (MIST), are observed via blood-oxygenation-level-dependent functional magnetic resonance imaging (BOLD fMRI) and simultaneous positron emission tomography (PET) imaging using the radiotracer 18 Fluor (18F)-N,N-diethyl-2-[4-(2-fluoroethoxy)phenyl]-5,7-dimethylpyrazole[1,5-a]pyrimidine-3-acetamide (DPA)-714, which targets the 18 kilodalton (kDA) translocator protein (TSPO) of activated microglia. Every participant will receive 0.4 ng/kg body weight of LPS and saline on separate treatment visits, separated by a 2-3 months wash-out period.

ELIGIBILITY:
Inclusion Criteria:

* Male
* Healthy
* Age 18-45 years
* BMI 18.5-25 kg/m2
* Proficient in English and/or Dutch

Exclusion Criteria:

* Have previous or current neuropsychiatric disorders or have history of major head trauma
* Have any disorder, which in the Investigator's opinion might jeopardise your safety or compliance with the study
* Have any prior or current treatment(s) that might jeopardise your safety or that would compromise the integrity of the study
* Have any prior and recent medication use (especially antibiotics, cardiovascular drugs, steroids, non-steroid anti-inflammatory drugs, centrally effective drugs)
* Are participating in an interventional Trial with an investigational medicinal product (IMP) or device
* Have current or previous infection or vaccination within the last 8 weeks
* Have pathological values of blood indices and certain genetic profiles that will affect brain imaging results (we will conduct a blood screening before starting the study)
* Had strong physical activity (e.g. swimming, football, running more than 8 km per hour, carrying heavy loads) 24h before the start of the experiment.
* Are a smoker
* Are a night-shift worker
* Have recent or previous use of psychotropics within the last year
* Have regular high alcohol use (>4 drinks/week)
* Have any brain imaging contraindications:

  * Have claustrophobia or too much uneasiness in limited spaces (in order to tolerate confinement during the scanning procedures).
  * Have severe back problems that will interfere with lying on your back in the scanner with no movement for long durations.
  * Have any condition that would interfere with MRI studies (e.g., cochlear implant, metal fragments in eyes, cardiac pacemaker, neural stimulator, and metallic body inclusion or other metal implanted in the body). To check this, you will need to fill out a checklist before the procedure.
* You and/or your partner is planning to become pregnant during and up to one month of the completion of the study

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-05-03 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Blood-oxygenation-level-dependent functional magnetic resonance imaging (BOLD fMRI) response to acute stress task | 2 hours after the single i.v bolus administration of LPS or saline
  BOLD fMRI responses to the Montreal Imaging Stress Task (MIST) after administration of LPS compared to saline
Binding potential of [18F]-DPA-714 radiotracer | 2 hours after the single i.v bolus administration of LPS or saline
  The change in [18F]-DPA-714 binding potential with and without LPS administration (%∆BPND)

SECONDARY OUTCOMES:
Concentration of serum cytokines | From 1 hour prior to intervention to 6 hours post-intervention
  Serum samples will be used for the quantification of inflammatory cytokines tumor necrosis factor alpha (TNF-α), interleukin-1β (IL-1β), interferon-γ (IFN-γ), IL-6, IL-8, IL-1 receptor agonist (RA), IL-4, and IL-10 using the Meso Scale Discovery (MSD) electrochemiluminescence validated (V-PLEX) system.
Concentration of serum C-reactive protein (CRP) | From 1 hour prior to intervention to 24 hours post-intervention
  Serum samples will be used to analyze high sensitive CRP (hs-CRP) levels using latex-enhanced immunonephelometric test.
Concentration of serum free cortisol | From 1 hour prior to intervention to 24 hours post-intervention
  Serum samples will be used to analyze the concentration of free cortisol in the circulation using electrochemiluminescence.
Concentration of plasma Adrenocorticotropic Hormone (ACTH) | From 1 hour prior to intervention to 24 hours post-intervention
  Plasma samples will be used to analyze the concentration of ACTH in the circulation using electrochemiluminescence.
Pulse rate | From 1 hour prior to intervention to 6 hours post-intervention
  To monitor the participants' condition and response to the treatment, pulse rate will be recorded every hour. Pulse rate will be measured using a pulse oximeter and/or digital sphygmomanometer and recorded in beats per minute.
Systolic blood pressure | From 1 hour prior to intervention to 6 hours post-intervention
  To monitor the participants' condition and response to the treatment, systolic blood pressure will be recorded every hour. Systolic blood pressure will be measured using a digital sphygmomanometer and recorded in millimeters of mercury (mmHg).
Diastolic blood pressure | From 1 hour prior to intervention to 6 hours post-intervention
  To monitor the participants' condition and response to the treatment, diastolic blood pressure will be recorded every hour. Diastolic blood pressure will be measured using a digital sphygmomanometer and recorded in millimeters of mercury (mmHg).
Body temperature | From 1 hour prior to intervention to 6 hours post-intervention
  To monitor the participants' condition and response to the treatment, body temperature will be recorded every hour. Temperature will be taken in the ear using a tympanic thermometer and recorded in degrees of Celsius (°C).
Scoring of the Generic Assessment of Side Effects (GASE) questionnaire | From 1 hour prior to intervention to 7 days post-intervention
  General side effects will be assessed and recorded in a structured, validated approach using the Generic Assessment of Side Effects (GASE). The GASE consists of 36 items asking for most frequently reported side effects for drugs based on the FDA adverse event reporting system database from all countries. Symptoms of all body parts during the last seven days will be self-reported and rated based on severity from 0 (not present) to 3 (severe).
Scoring of the Sickness Questionnaire (SicknessQ) | From 1 hour prior to intervention to 24 hours post-intervention
  To comprehensively measure sickness behaviour during the test day, the Sickness Questionnaire (SicknessQ) will be used. The SicknessQ is a brief and psychometrically sound assessment instrument to measure perceived sickness behaviour. It is sensitive to LPS challenge and was developed based on acute sickness response to LPS endotoxemia in healthy individuals. The SicknessQ score was significantly increased by LPS challenge compared to placebo at 1.5 hours post-injection and subsided to non-significant levels after 4.5 hours. In addition, the increase in SicknessQ score was partly mediated by the relative increase in inflammatory cytokines.
Scoring of the State-Trait Anxiety Inventory, State Anxiety subscale (STAI-S) | From 1 hour prior to intervention to 24 hours post-intervention
  To measure momentary anxiety during the test day, the STAI-S will be used. This inventory is part of the State-Trait Anxiety Inventory (STAI). The STAI is a psychological inventory that measures two types of anxiety - state anxiety and trait anxiety. State anxiety is anxiety about an event, while trait anxiety is the level of anxiety related to an individual's character. The inventory consists of 40 questions, with 20 questions specifically for state anxiety, rated on a 4-point scale. State anxiety is rated with anxiety absent and anxiety present questions. Anxiety absent questions constitute the absence of anxiety in a statement like, "I feel secure." Anxiety present questions represent the presence of anxiety in a statement like "I feel worried." The 4-point scale are as follows: 1 'not at all', 2 'somewhat', 3 'moderately so', and 4 'very much so'.
Scoring of the State-Trait-Anxiety and Depression Scale (STADI) | From 1 hour prior to intervention to 24 hours post-intervention
  The State-Trait Anxiety-Depression Inventory aims to recognize and differentiate symptoms of anxiety and depression. It consists of 40 self-report items that distinguish between temporary (state) and chronic conditions (trait). The rating scale consists of a 4-point Likert-type scale ranging from 1 (not at all) to 4 (very much). The STADI has a 4-factor structure of anxiety and depression including emotionality, worry, dysthymia, and anhedonia.
Scoring of the Stanford Sleepiness Scale (SSS) | From 1 hour prior to intervention to 24 hours post-intervention
  The Stanford Sleepiness Scale (SSS) is a self-report questionnaire that aims to quickly assess the levels of sleepiness throughout the day and track overall alertness at each hour of the day. It is commonly used in research and clinical settings to assess the effectiveness of a specific treatment. The scale is rated from 1 to 7 with 1 being wide awake and 7 being sleep onset. A rate of X is given if the respondent is asleep.
Scoring of the Positive and Negative Affect Schedule (PANAS) | From 1 hour prior to intervention to 24 hours post-intervention
  The PANAS consists of two 10-item mood scales and was developed to provide brief measures of negative affect (NA) and positive affect (PA). NA and PA reflect dispositional dimensions, with high-NA epitomized by subjective distress and unpleasurable engagement, and low-NA by the absence of these feelings. By contrast, PA represents the extent to which an individual experiences pleasurable engagement with the environment. Thus, emotions such as enthusiasm and alertness are indicative of high-PA, whilst lethargy and sadness characterize low-PA. Respondents are asked to rate the extent to which they have experienced each particular emotion within a specified time period, on a 5-point scale. The scale points are: 1 'very slightly or not at all', 2 'a little', 3 'moderately', 4 'quite a bit', and 5 'very much'.
Scoring of the Multidimensional Mood Questionnaire (MDMQ) | From 1 hour prior to intervention to 24 hours post-intervention
  The MDMQ is a well-validated 24-item questionnaire commonly used to quickly evaluate the mental state and mood of a respondent. It consists of 24 items to measure three current psychological states in bipolar dimensions of: good vs. bad, awake vs. tired, and calm vs. nervous. Each item is rated with a 5-point rating scale. The results range between 1 (feeling bad, tired, nervous) and 40 points (feeling good, awake, calm) for each dimension, summing up to an overall maximum count of 120 points (maximum scores for feeling good, awake, and calm) for the whole questionnaire.

OTHER OUTCOMES:
Concentration of serum short-chain fatty acids (SCFAs) | From 1 hour prior to intervention to 6 hours post-intervention
  Serum blood will be used to quantify SCFA levels using gas chromatography/mass spectrometry (GC-MS) for exploratory analysis.
Quantitative profile of microbiota | On each intervention/placebo day
  Quantitative microbiota profiling will be performed using metagenomic shotgun sequencing and/or 16s sequencing for exploratory analysis.
Scoring of the Bristol Stool Score (BSS) | On each intervention/placebo day
  Self-report of the Bristol Stool Score will be recorded to determine fecal consistency for exploratory analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Lukas Van Oudenhove, MD, PhD, Principal Investigator — KU Leuven; Kristin Verbeke, Pharm, PhD, Principal Investigator — KU Leuven; Boushra Dalile, PhD, Principal Investigator — KU Leuven
Locations (1):
- UZ/KU Leuven, Leuven, Flemish Brabant, Belgium

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data (IPD) that underlie results in a publication will be made available to other researchers with all identifying information removed.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: The data will become available upon publication with no time limitations.
Access Criteria: The data will be publicly available.